CLINICAL TRIAL: NCT06828419
Title: A Clinical Study on the Feasibility and Safety of Abdominal Endoscopic Single-port Surgery System to Assist Gynecological Day Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SAHoWMU-CR2024-07-124
Record Dates: First submitted 2025-02-04; First posted 2025-02-14 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Adenopathy; Uterine Fibroids; Ovarian Cysts; Adnexal Mass; Ovarian Diseases; Adnexal Cyst; Adnexal Diseases
Keywords: robotic-assisted laparoscopic single-site surgery (R-LESS); single-port robot system (SPRS); day surgery
MeSH Terms: conditions — Lymphadenopathy; Leiomyoma; Ovarian Cysts; Ovarian Diseases; Adnexal Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Domestic single-port laparoscopic surgery system group (Other): The domestic single-port robotic laparoscopic surgery system is a new minimally invasive surgical method. Compared with traditional laparoscopic surgery, it establishes the surgical approach through the natural scar umbilicus of the human body, thus bringing less trauma and beautiful experience to patients
  Interventions: Device: Domestic single-port laparoscopic surgery system

INTERVENTIONS:
Device: Domestic single-port laparoscopic surgery system — The minimum distance of the single-port surgical system from the port is 5-7cm to obtain the instrument bending space. The load capacity of surgical tools is increased from 2N to 5N, which greatly improves the structural reliability. At the same time, it can realize 6 degrees of freedom movement。

SUMMARY:
In this study, a prospective study is used to select patients who will undergo intra-abdominal endoscopic single-port surgery system for benign gynecological diseases from February 2025 to December 2026 in the Second Affiliated Hospital of Wenzhou Medical University, including hysterectomy, myomectomy, ovarian cyst removal and adnexectomy. The study will perform statistical analysis to evaluate the feasibility and the main factors affecting the safety of intra-abdominal endoscopic single-port surgery system(SR-ENS-600) used in gynecological day surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Women aged 18 to 75 years old, with a body mass index (BMI) of no more than 32 kg/m2;
2. Conscious, no history of mental illness, accompanied by an adult during the perioperative period;
3. Educate the subjects, who are willing to undergo day surgery, understand and accept the surgical method and anesthesia method;
4. Subjects and families understand perioperative care and are willing and able to complete post-discharge care;
5. Elective surgery, no serious complications affecting the operation and prognosis, aCCI age adjusted comorbidity index 0 points;
6. According to the adhesion risk scoring system of European Anti-Adhesions in Gynaecology Expert Panel (ANGEL), the adhesion risk was divided into three levels: high, medium and low. Subjects with low risk (0 to 12 points) and abdominal wall scarring and pelvic cavity B-ultrasonography do not indicate obvious pelvic cavity adhesion wiil be included.

Exclusion Criteria:

1. Moderate and high-risk patients will be excluded based on ANGEL adhesion risk scoring system;
2. Subjects with hemorrhagic rupture of ectopic pregnancy and unstable vital signs;
3. Genital tract infection or in the acute phase of systemic infection;
4. Subjects on long-term anticoagulant therapy or with coagulation dysfunction;
5. Subjects have severe heart and lung disease, liver and kidney dysfunction, and cannot tolerate anesthesia;
6. A history of abdominal or diaphragmatic hernia, abnormal umbilical cord development, or umbilical surgery;
7. Not willing to undergo endoscopic surgery;
8. Participated in other drug and device clinical trials within 3 months before surgery.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Estimated)
Dates: Start 2025-04-10 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Day Surgery Success Rate | Patient recruitment ends and all patients complete surgery, up to 2 years
  Day surgery success rate means that no other operation is performed during the operation and the patient is discharged within 48 hours.

SECONDARY OUTCOMES:
Time of Operation | From pre-surgery to the end of surgery，up to 12 hours
  Time of operation includes total operation time, operator teleoperation time, robot system parking time and instrument docking time。
Blood Loss Evaluation | From the time of hemoglobin measurement before surgery to the time of hemoglobin measurement after surgery, up to 1 day after surgery
  The estimated intraoperative blood loss and the difference of hemoglobin before and after operation.
Surgeon Satisfaction Evaluation | Up to 1 day after surgery
  Surgeon satisfaction questionnaire
Time of First Postoperative Anal Exhaust | Up to 2 day after surgery
  time recording
First Spontaneous Urination Time | Up to 2 day after surgery
  Time recording
Pain Score | 4 hours after surgery
  Visual Analogue Scale(VAS)
Hospital Stays | From the date of admission to the Date of discharge, assessed up to 2 days
  Time
Postoperative Rehabilitation Evaluation | Within 1 day after surgery; 24 hours and 30 days after discharge
  Quality of Life-15(QOL-15)
Abdominal Incision Healing | Within 1 day after surgery
  Observation
Scar Satisfaction | 30 days after discharge
  Scar Cosmesis Assessment and Rating(SCAR)
Discharge Assessment | Within 1 day after surgery, 4 hours after discharge
  Postanesthesia Discharge Score(PADS)
Postoperative Complication | 4 hours, 24 hours and 30 days after discharge
  Telephone, Wechat official account and outpatient follow-up
Quality and Safety Evaluation of Day Surgery | 30 days after discharge
  13 indexes of quality and safety evaluation of day surgery
Safety Evaluation | Day of surgery and within 1 day after surgery; 4 hours, 24 hours and 30 days after discharge
  6 indexes of safety evaluations

CONTACTS AND LOCATIONS:
Locations (1):
- Second Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan: Study Protocol (2025-02-22): https://cdn.clinicaltrials.gov/large-docs/19/NCT06828419/Prot_SAP_002.pdf
  • Study Protocol and Informed Consent Form: Informed Consent Form (2025-02-22): https://cdn.clinicaltrials.gov/large-docs/19/NCT06828419/Prot_ICF_003.pdf
  • Informed Consent Form: New Technology and New Project Informed Consent Form (2024-04-26): https://cdn.clinicaltrials.gov/large-docs/19/NCT06828419/ICF_004.pdf